CLINICAL TRIAL: NCT05965440
Title: Impact of Dapagliflozin on Intestinal Microbiota Composition and on the Metabolites Derived from the Intestinal Microbiota in Non-diabetic Chronic Renal Failure Patients
Acronym: DAPA-GUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL23_0410
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Diseases
Keywords: CKD; gliflozine; gut microbiota; metabolomic; uremic toxin
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- impact of Dapagliflozin on Intestinal Microbiota on chronic renal failure patients (Other): * Addition of 3 blood tubes of 5mL during the collection for the treatment
  * Collection of fresh urine (7 mL)
  * Collection of stools by the participant at his home
  * Collection of fresh stools for patients participating in the ancillary study
  * Constitution of a biocollection (blood, urine and stool)
  * Food collection for 3 days with no impact on patient follow-up
  * Stool appearance sheet to be completed by the patient at each collection
  Interventions: Drug: impact of Dapagliflozin on Intestinal Microbiota on chronic renal failure patients

INTERVENTIONS:
Drug: impact of Dapagliflozin on Intestinal Microbiota on chronic renal failure patients — Analysis of microbiota

SUMMARY:
Chronic kidney disease (CKD) is a common disease affecting 10-12% of the adult population and characterize with high-risk cardiovascular morbidity and mortality with progression of CKD. Treatment with sodium-glucose cotransporter 2 inhibitors (iSGLT2) not only improves hyperglycemia and type 2 diabetes (T2D) but also results in body-weight loss, a reduction in blood pressure, and a decrease of cardiovascular events and progression of renal failure in both diabetes and non-diabetes patients.(Heerspink et al. 2020) Therefore, dapagliflozin is now associated with the inhibitors of the renin-angiotensin system to reduce kidney events.

However, the mechanisms underlying the effects of dapagliflozin on the renal function remain unclear. When renal failure occurs, it impairs the removal of several metabolites called uremic retention solutes. If these retention solutes exhibit deleterious interferences with biochemical/physiological functions, they are referred to as uremic toxins as they can contribute to the manifestations of the uremic syndrome and are associated with a high cardiovascular morbidity and mortality and with progression of CKD. Many of the uremic toxins are not produced by the body itself but rather derived from gut microbiota metabolism such as the well-known trimethylamine-N-oxide (TMAO),p-cresyl sulfate (PCS), phenyl sulfate (PS), indoxyl sulfate (IS), and indole-3-acetic acid (IAA).The gut microbiota composition in a uremic context has been the subject of an increasing number of publications and majority of them confirm a decrease of gut microbiota richness and deep modifications.Recently, an animal study suggested that dapagliflozin, subtly improve the composition of the gut microbiota in mice with T2D and another preliminary clinical study didn't observe a modification in the fecal microbiome after dapagliflozin initiation.But in other study, empagliflozin significantly reshaped the gut microbiota after 1 month of treatment in T2D patients and be associated with shifts in plasma metabolites. Similarly, canagliflozin reduces plasma uremic toxins in a CKD mice model.However, it remains unknown whether treatment with dapagliflozin alters the gut microbiota in CKD patients without T2D; furthermore, the relationship between the gut microbiota, uremic toxins production and CKD-related beneficial effects of dapagliflozin remains elusive.

Herein, the investigator will investigate the clinical benefits of dapagliflozin and possible associations between its renal function benefits and alterations in plasmatic gut microbiota-derived metabolites and the gut microbiota composition in non-T2D CKD patients. To this end, the investigator will conduct an observational clinical trial in non-T2D CKD patients with the primary aim of investigating dapagliflozin-induced compositional changes of intestinal gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old
* Non-diabetic patient
* PChronic renal failure patient with a medical indication for the introduction of dapagliflozin as part of routine care: o either according to the marketing authorization, namely:

  * A GFR estimated between 25 and 60 mL/min/1.73m2 according to the CKD EPI formula.
  * A urinary albumin/creatinine ratio > 200mg/g and < 5000 mg/g
  * Be treated with the maximum tolerated dose of renin-angiotensin system inhibitors for at least 4 weeks. o or according to the nephrologist's assessment if the patient has other indications such as chronic heart failure according to the marketing authorization or any patient with a GFR > 20 ml/min according to the KDIGO recommendations for the management of CKD
* BMI between 18 and 30 kg/m2
* Patient not taking dapagliflozin (or any other treatment containing iSGLT2 or iSGLT1)
* Very regular bowel movements between 24 and 48 hours
* Patient following the dietary recommendations recommended during CKD (a sodium intake targeting 6g NaCl/day +/-20% and a protein intake of 0.6g/kg/d +/-20%)
* Affiliation to social security

Exclusion Criteria:

* Taking drugs can interfere with the intestinal microbiota (prebiotics, probiotics, postbiotics, antibiotics) in the last 6 weeks
* Patient using high dose laxatives (more than 2 per day, for more than 3 months)
* Patient with a foreseeable transplant or dialysis project within the next 6 months.
* Patient with a colectomy, a resection of the small intestine or a cholecystectomy
* Patient with a progressive and unstabilized inflammatory, infectious, cardiovascular or neoplastic disease
* Inability to understand the nature, follow-up and possible consequences of the study.
* Patient in exclusion period from previous study or already participating in a clinical research protocol having an impact on the endpoints of the study
* Patient under guardianship or in safeguard of justice
* Pregnant, parturient or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity and beta diversity size of the intestinal microbiota after 12 weeks of daily treatment with dapagliflozin compared to alfa and beta diversity size before initiation of treatment. | Before and 12 weeks after initiation of treatment with dapagliflozin
  The analysis of the microbiota by 16s sequencing of bacterial DNA will be carried out on the GenEPII platform located at the Croix Rousse hospital, Hospices Civils de Lyon (Pr Sophie JARRAUD).

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology department, Hôpital Lyon Sud, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No